CLINICAL TRIAL: NCT03207789
Title: Prospective Collection of Data in Patients With T-cell Lymphomas Distributed in the Five Distinct Macro Regions of Brazil
Brief Title: T-cell Brazil: Prospective Collection of Data in T-cell Lymphomas Patients
Acronym: Tcell-Brazil
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: CAAE: 69605517.1.1001.5487
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: T-cell Lymphoma; NK-Cell Lymphoma; T-cell Lymphoma Adults
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The designed study follows up on the previous one by the international T-cell project (Bellei et al,, 2012) and its purpose is to verify whether a prospective collection of data would permit access to more accurate information permitting a better definition of prognosis and investigation of more adequate treatment strategies for these neoplasms.

The analysis of patients distributed in all five macro regions of the country and a comparison among them will provide a real picture of the disease in Brazil, limiting the bias probably found in the previous projects.

DETAILED DESCRIPTION:
Patients with diagnosis histologically confirmed T-cell or NK-cell lymphoma will be registered in the study, despite of their planned treatment. Registration will be made on-line on a key restricted accessible web-database after obtaining the informed consent dated and signed by the patient. Every registered patient has as well to undergo a central histopathology review by a panel of experts. The referring pathologist will collect and review the patological material sent by the participating centers, without knowing the clinical outcome of the patient. Validated cases have to be supplied of information regarding treatment procedures and follow up updating for at least 5 years. The primary endpoint is the overall survival and other endpoints such as event free survival; progression free survival, complete and partial response rates.

ELIGIBILITY:
Inclusion Criteria:

* Dated and signed informed consent;
* T-cell or NK-cell diagnosis;
* Tissue biopsies adequate for diagnosis and classification and available for centralized review;
* clinical, laboratory, image data available and registred in the website.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed histologically diagnosis of T-cell or NH-cell lymphoma in any of 5 macro region of Brazil
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis during the first year of T-cell Brazil Registry | 12 months of registring
  Descriptive analysis and Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Eliana CM Miranda, M.Ed.; Ph.D., Study Chair — Grupo de Estudos Multicentricos em Onco-Hematologia

IPD SHARING:
Plan to Share IPD: No